CLINICAL TRIAL: NCT03817346
Title: A Phase I, Randomised, Double-blind, Placebo-controlled Study in Healthy Male Volunteers to Investigate the Safety, Tolerability and Pharmacokinetics of Ascending Single Oral Doses of GT-002
Brief Title: Study of Ascending Single Oral Dose of GT-002 in Healthy Volunteers
Acronym: GAB-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gabather AB (Industry)
Collaborators: Smerud Medical Research International AS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: GAB-001
Record Dates: First submitted 2018-12-11; First posted 2019-01-25 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Safety and Tolerability
Keywords: Safety; Tolerability; Pharmacokinetics

STUDY DESIGN:
Intervention Model Description: Single ascending dose
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blinde
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental GT-002 SAD (Active Comparator): Healthy volunteers meeting eligibility criteria will be sequentially randomized to each dose cohort (up to 7 dose ascending cohorts) to receive either GT-002 or placebo. The study drug (GT-002 or placebo) will be administered orally as a single dose. Six of out 8 subjects per cohort will be randomized to receive GT-002.
  Interventions: Drug: GT-002
- Experimental Placebo oral capsule SAD (Placebo Comparator): Healthy volunteers meeting eligibility criteria will be sequentially randomized to each dose cohort (up to 7 dose ascending cohorts) to receive either GT-002 or placebo. The study drug (GT-002 or placebo) will be administered orally as a single dose. Two of out 8 subjects per cohort will be randomized to receive GT-002.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: GT-002 — Single ascending dose
  Arms: Experimental GT-002 SAD
Drug: Placebo oral capsule — Comparator single ascending dose
  Arms: Experimental Placebo oral capsule SAD

SUMMARY:
This study does not target any disease or condition in itself, but is evaluating the safety, tolerability and pharmacokinetics of single oral doses of GT-002 in the setting of healthy volunteers.

A longer-term objective is to apply the findings from this study to design and later conduct a clinical development programme of GT-002 as a medication to treat schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing and able to give written informed consent for participation in the study. Sufficient command of the Finnish language will be needed for informed consent and adequate communication with the study personnel.
2. Healthy male subjects from 18 up to 45 years of age.
3. Body mass index (BMI) from 18 kg/m2 up to 28 kg/m2.
4. Body weight from 60 kg up to 120 kg.
5. Clinically normal medical history, physical findings, vital signs, ECG and laboratory values as judged by the investigator at the time of the screening visit. A subject with a clinical abnormality or laboratory parameters outside of the reference range for the population being studied may be included at the investigator´s discretion provided the finding is unlikely to introduce additional risk factors, jeopardize study integrity, or to interfere with the study assessments or procedures.
6. Subjects must be willing to use condom or other contraceptive methods with a failure rate of < 1% and refrain from donating sperm from the date of dosing until one month after last dosing.

   -

Exclusion Criteria:

1. Current or history of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
2. History of any type of cancer.
3. Subjects considered unlikely to comply with study procedures, restrictions and requirements
4. Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the administration of investigational product that is likely to introduce additional risk factors, jeopardize study integrity, or to interfere with the study assessments or procedures
5. Any clinically significant abnormalities in clinical chemistry, haematology, coagulation or urinalysis results at the time of screening visit as judged by the investigator
6. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody or human immunodeficiency virus (HIV)
7. After 10 minutes of supine rest, abnormal vital signs defined as any of the following:

   1. Systolic blood pressure > 140 mm Hg (average of two measurements)
   2. Diastolic blood pressure > 90 mm Hg (average of two measurements)
   3. Heart rate < 40 or > 85 beats per minute (average of two measurements)
   4. Body temperature (auricular) ≥38oC
8. Prolonged QTcF interval (>450 ms), clinically significant cardiac arrhythmia or any other clinically significant abnormalities in the resting ECG as judged by the investigator
9. Intake of any medication, vitamin or mineral supplement product that could affect the outcome of the study, within 2 weeks prior to the first study treatment administration or less than 5 times the half-life of the medication. Possible prior use of enzyme inducing drugs will be considered case-by-case by the investigator.
10. Any blood donation/blood loss > 250 ml during the 3 months prior to screening
11. Has received another new chemical entity (defined as a compound which has not been approved for marketing) or has participated in any other clinical trial that included drug treatment within 3 months of the administration of investigational product in this study. Subjects consented and screened but not dosed in previous phase I studies can be included in this study.
12. Current or history of alcohol or drug abuse within the last 5 years, current excessive use of alcohol (current regular alcohol drinking of more than 24 units/week) or use of illicit drugs.
13. Positive screen for drugs of abuse at screening or on admission to the unit or positive breath test result for alcohol at screening or on admission to the unit prior to the administration of investigational product.
14. Known allergy to the components used in the formulation of GT-002.
15. Current smokers or users of nicotine products. Irregular use of nicotine (e.g. smoking, snuffing, and chewing tobacco) up to five doses per week is allowed before screening visit.
16. Intake of >5 cups of coffee/day or the corresponding amount of other caffeine containing beverages (e.g. energy drinks containing caffeine) during the study.
17. Subjects who have planned any scheduled invasive treatment or medical/surgical procedure during the study period.

    -

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 32 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Day 1 to day 3
  To evaluate the safety and tolerability GT-002 in healthy subjects by assessing the number, severity and type of adverse events, including changes in vital signs, physical examinations, laboratory safety tests and ECGs

SECONDARY OUTCOMES:
Pharmacokinetic parameter AUCt | Day1 to day 3
  Area under the curve from the time of dosing until the last quantifiable concentration
Pharmacokinetic parameter AUC0-24 | Day1 to day 2
  Area under the curve from the time of dosing until 24 hours post dosing
Pharmacokinetic parameter AUC0-infinity | day 1 to day 3
  Area under the curve from the time of dosing extrapolated to infinity
Pharmacokinetic parameter Cmax | Day 1 to day 3
  Maximum concentration (Cmax)
tmax | Day 1 to day 3
  Time to maximum concentration
t1/2 | Day 1 to day 3
  Apparent terminal elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Peltonen, Study Chair — Smerud Medical Research Finland Ab/Oy
Locations (1):
- CRST Oy, Clinical Research Services Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: No